CLINICAL TRIAL: NCT01796054
Title: Effectiveness of a Mind-body Stress Reduction Program for Nurses: A Randomized Controlled Study
Brief Title: Stress Free Now, a Mind-body Reduction Program for Nurses
Acronym: SFN-Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-1398
Record Dates: First submitted 2013-02-15; First posted 2013-02-21 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Psychological Stress; Anxiety; Depression
Keywords: Perceived stress; Burnout; Mindfulness; Intent to leave nursing
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stress Free Now with group support (Experimental): Randomized participants have access to online stress reduction program, Stress Free Now. Participants will log in to online program, read daily lessons and practice therapeutic exercises. They will also attend weekly group support session during 6-week program
  Interventions: Behavioral: Stress Free Now online program; Behavioral: Group support session
- Stress Free Now (Experimental): Randomized participants have access to online stress reduction program, Stress Free Now, for 6 weeks. Participants will log into online program, read daily lessons and practice therapeutic exercises.
  Interventions: Behavioral: Stress Free Now online program
- Control (No Intervention): Randomized participants do not have access to online stress reduction program, Stress Free Now, nor do they attend weekly group support sessions.

INTERVENTIONS:
Behavioral: Stress Free Now online program — Stress Free Now is an online stress reduction program. Participants will log into online program, read and practice daily and weekly activities.
  Arms: Stress Free Now; Stress Free Now with group support
Behavioral: Group support session — Participants will meet weekly for group support session to review online lessons and relaxation therapies.
  Arms: Stress Free Now with group support

SUMMARY:
Mindful meditation sessions have been associated with an improvement in mindfulness, perceived stress, psychological well-being, anxiety, hostility, and depression. Meditation has been associated with a decrease in autonomic sympathetic activity, heart rate, oxygen consumption and energy expenditure. Randomized controlled trials of online mindfulness and relaxation programs have been studied in patients with conditions such as irritable bowel syndrome, headache, depression, fibromyalgia, and insomnia. Nurses may benefit from such programs given levels of job stress. This study will determine whether an online stress reduction program that incorporates meditation with and without concomitant group support reduces burnout among nurses, including emotional exhaustion and depersonalization. The proposed research study will utilize Stress Free Now, an online stress reduction program developed by Cleveland Clinic Wellness Institute.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-center research study of an online intervention with peer group support to reduce stress in nurses. All participants will be assigned to the intervention or control groups by random number allocation. The duration of the intervention is 6 weeks; follow-up is at 6 and 24 weeks; the duration of the study is 6 months (24 weeks). Total individual participant time commitment will depend on particular intervention or control group assignment. Both intervention and control groups will be requested to complete a set of questionnaires at weeks 0, 6, and 24. The questionnaires will take an estimated 45 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* work as a full-time or part-time nurse at Cleveland Clinic
* have regular internet and email access and be willing and able to attend group support sessions
* work at least one weekday during the week in order to attend orientation and/or group support sessions

Exclusion Criteria:

* participating in another stress reduction research study
* pregnant, lactating, or planning to be pregnant in the next 6 months
* hospitalized for depression in past 12 months
* vacation time away from work for more than 1 week during the first 2 months of the study
* current diagnosis of schizophrenia, other psychotic or bipolar disorder
* other medial, psychiatric, or behavioral limitations that may interfere with study participation or the ability to follow the intervention protocol
* unwilling or uninterested in participating in group sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Burnout | 24 weeks
  Measured by Maslach Burnout Inventory Human Services Survey

SECONDARY OUTCOMES:
Perceived stress | 24 weeks
  Measured by Perceived Stress Scale
Self-reported BMI | 24 weeks
Emotional well-being | 24 weeks
  Measured by RAND Short-Form (SF)-36
Insomnia | 24 weeks
Psychosomatic symptoms | 24 weeks
  Measured by Psychosomatic Symptoms Checklist
Mindfulness | 24 weeks
  Measured by Five Factor Mindfulness Questionnaire
Intent to leave nursing | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bernstein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States